CLINICAL TRIAL: NCT02493556
Title: Effect of Low-level Laser Therapy on Exercise-induced Muscle Damage: a Randomized Clinical Trial
Brief Title: Effect of Low-level Laser Therapy on Exercise-induced Muscle Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Bruno Manfredini Baroni, Phd, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 38076514.0.0000.5345
Record Dates: First submitted 2015-07-07; First posted 2015-07-09 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-07

CONDITIONS: Muscle Damage
Keywords: Phototherapy; Plyometric exercise; Muscle recovery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- LLLT before muscle damage (Experimental): Low Level Laser Therapy (LLLT) will be applied before the exercise protocol on one lower limb, while the other will receive placebo treatment. Phototherapy will be applied with an equipment of 810nm and a cluster with five diodes on eight different points of quadriceps muscle, totalizing a dosage of 240J.
  Interventions: Device: LLLT before muscle damage
- Placebo LLLT before muscle damage (Placebo Comparator): Placebo LLLT will be applied before the exercise protocol on one lower limb, while the other will receive real treatment. Placebo treatment will also be applied on eight different points of quadriceps muscle, but the equipment will be turned off.
  Interventions: Device: Placebo LLLT before muscle damage
- LLLT after muscle damage (Active Comparator): Low Level Laser Therapy (LLLT) will be applied after the exercise protocol on one lower limb, while the other will receive placebo treatment. Phototherapy will be applied with an equipment of 810nm and a cluster with five diodes on eight different points of quadriceps muscle, totalizing a dosage of 240J.
  Interventions: Device: LLLT after muscle damage
- Placebo LLLT after muscle damage (Placebo Comparator): Placebo LLLT will be applied after the exercise protocol on one lower limb, while the other will receive real treatment. Placebo treatment will also be applied on eight different points of quadriceps muscle, but the equipment will be turned off.
  Interventions: Device: Placebo LLLT after muscle damage

INTERVENTIONS:
Device: LLLT before muscle damage
  Arms: LLLT before muscle damage
Device: Placebo LLLT before muscle damage
  Arms: Placebo LLLT before muscle damage
Device: LLLT after muscle damage
  Arms: LLLT after muscle damage
Device: Placebo LLLT after muscle damage
  Arms: Placebo LLLT after muscle damage

SUMMARY:
Introduction: The effects of Low Level Laser Therapy (LLLT) on exercise-induced muscular damage have been studied over the last years. Studies have been conducted on animals and humans in order to try to show the benefits of the intervention, but there is still conflicting evidence about its protective and therapeutic effects.

Objectives: To describe the effects of LLLT on pain, strength and muscular inflammation after plyometric exercise.

Methods: A randomized, double-blinded, placebo-controlled trial with participation of 20 male healthy volunteers will be performed. Healthy and physically active individuals, aged between 18 and 35 years, with no history of injury on the lower limbs or contra-indications to maximal exercise performance will be included. A protocol of 10 series with 10 repetitions of the countermovement jump will be used to induce muscle damage at the lower limbs. Immediately before or after the exercise protocol, LLLT will be applied on one lower limb, while the other will receive placebo treatment. Phototherapy will be applied with an equipment of 810nm and a cluster with 5 diodes on 8 different points of the knee extensor muscle, totalizing a dosage of 240J. The placebo treatment will be held on the same way, but the equipment will be turned off. The volunteers will be evaluated at baseline (before the exercise protocol) and at follow-up of 24, 48 and 72 hours. The following outcomes will be evaluated: knee extensors isometric peak torque by Isokinetic Dynamometer, pain by Visual Analogue Scale and muscular tissue echo intensity by Ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged between 18 and 35 years;
* Sedentary or physically active individuals who exercise up to 3 times per week.

Exclusion Criteria:

* Individuals who participate in systematic exercise training;
* Individuals who participate in strength training for the lower limbs;
* Individuals with lower or upper limb injuries;
* Individuals with contra-indications to maximal exercise performance (due to neurological, cardiovascular or respiratory conditions);
* Individuals who show difficulties to understand the study protocol.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Knee extensors isometric peak torque (Nm) | Baseline and 24, 48 and 72 hours follow-up
  Isokinetic Dynamometer

SECONDARY OUTCOMES:
Knee extensors soreness (Visual Analogue scale) | Baseline and 24, 48 and 72 hours follow-up
Knee extensors echo intensity (number of white and black pixels) | Baseline and 24, 48 and 72 hours follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Baroni, phD, Study Director — Federal University of Health Science of Porto Alegre
Locations (1):
- Federal University of Health Science of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil